CLINICAL TRIAL: NCT00299845
Title: Randomized Trial for Pharmacogenomics-based Proton Pump Inhibitor Therapy in Children
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Osaka University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG-ped-LPZ-01
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2006-09

CONDITIONS: Gastroesophageal Reflux
Keywords: gastroesophageal reflux; children; lansoprazole; cytochrome P450 2C19 (CYP2C19); pharmacogenomics; genetic polymorphisms; individualized medicine; pharmacokinetics/dynamics
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole

SUMMARY:
Proton pump inhibitors are administered to children as off-label use in Japan. The purpose of this study is to evaluate the effects of CYP2C19 genotypes on pharmacokinetic /pharmacodynamic profiles of PPI in children. The results will provide the beneficial information for the individualized medicine of PPI in children.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastroesophageal reflux
* The patient's parent or guardian gives written informed consent including pharmacogenomic analysis
* The patient is willing and able to give assent to participate.

Exclusion Criteria:

* Serious hepatic disease, pulmonary disease, renal disease and blood disorder
* Inadequate clinical conditions

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Azuma, MD, Study Chair — Graduate School of Pharmaceutical Sciences, Osaka University
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan